CLINICAL TRIAL: NCT05485077
Title: Colorectal Cancer Screening Cohort Study in Shougang Community Population Based on Polygene Methylation Detection Technology
Brief Title: A Prospective Cohort Study on Colorectal Cancer Screening in Community Population
Status: Recruiting | Type: Observational
Sponsor: Singlera Genomics Inc. (Industry)
Collaborators: Peking University Shougang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KYS-2022007
Record Dates: First submitted 2022-07-26; First posted 2022-08-03 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
Keywords: ctDNA methylation; Community population screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive group: All the subjects who completed colorectal cancer polygene methylation test at baseline completed colonoscopy within 3 months. Colorectal cancer diagnosed by colonoscopy, adenoma or polyp lesions found after treatment will reach the end of the study. The tumor history of family members was tracked for patients who met the end point of the study. The positive subjects who did not reach the end point of the study underwent three center visits at 12, 36 and 60 months after enrollment respectively, including history taking, colonoscopy, FIT test and blood CEA test. Another telephone follow-up was conducted at 24 and 48 months, respectively.
- Negative group: The subjects who completed colorectal cancer polygene methylation test at baseline, and those with negative test results (n= 500, direct extraction method) completed colonoscopy within 3 months. The end points and follow-up were the same as those in the positive group. The negative group was compared with the positive group to observe the difference of negative predictive value and survival outcome.

SUMMARY:
This study will validate the real world results of polygene methylation detection in colorectal cancer in a large prospective community cohort. In this study, questionnaire survey and polygene methylation detection technology of colorectal cancer were used as preliminary screening methods, and colonoscopy was used as further validation examination method to screen colorectal cancer and precancerous lesions. The diagnosis and outcome of all lesions were based on colonoscopy and pathological examination.

DETAILED DESCRIPTION:
1. The informed consent signed by shougang Community will be completed in the baseline period: Colorectal cancer risk factors assessment questionnaire, medical history collection, fecal immunochemical (FIT), carcinoembryonic antigen (CEA) blood test and blood bowel cancer gene methylation detection, for colorectal cancer gene methylation detection results more positive subjects and the result of the negative part of the subjects (n = 500), within 3 months after receiving the results complete colonoscopy.
2. Follow-up at 1, 2, 3, 4, and 5 years after baseline included: ① Central follow-up at 1, 3, and 5 years: history collection, colonoscopy, FIT test, and CEA examination; ② Telephone follow-up at the 2nd and 4th years: medical history was collected; (3) Survival outcome registration was performed in the fifth year; Follow-up history was collected at 1, 2, 3, 4, and 5 years after completion of baseline, and survival outcomes were registered at 5 years.
3. During the follow-up, the subjects were confirmed to be diagnosed with colorectal cancer by evaluation (colorectal cancer was diagnosed by colonoscopy), and the subjects who were treated after polyps or adenomas were found during colonoscopy also reached the study endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Chronological age ≥40 years;
2. Full capacity for action;
3. After enrollment, the participants were able to complete the Colorectal Cancer Risk Factor Assessment Questionnaire and the annual follow-up interviews;
4. In the course of the study, the information related to tumor diagnosis in other hospitals can be timely fed back to the researchers;

Exclusion Criteria:

1. History of colorectal cancer and other malignant tumors;
2. Previous colorectal resection;
3. undergoing any cancer-related treatment;
4. Patients who have received major surgical treatment such as blood transfusion or transplantation within 3 months;
5. Participate in other interventional clinical investigators within 3 months;
6. Pregnant or lactating women;
7. Have autoimmune disease, hereditary disease, mental illness/disability, etc
8. Poor compliance, unable to complete the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18000 samples from Shougang community
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2022-07-09 (Actual); Primary Completion 2028-07-09 (Estimated); Study Completion 2028-07-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of polygene methylation detection in colorectal cancer | assessed up to 72 months
  To investigate the sensitivity and specificity of polygene methylation in the diagnosis of colorectal cancer in community population, and to evaluate its value as an auxiliary diagnosis
Negative predictive value and positive predictive value of polygene methylation in colorectal cancer | assessed up to 72 months
  To obtain the positive predictive value and negative predictive value of polygene methylation test for colorectal cancer early screening, and compare with FIT test and blood CEA test.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, Doctor, Principal Investigator — Singlera Genomics Inc.
Locations (1):
- Peking University Shougang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schlemper RJ, Riddell RH, Kato Y, Borchard F, Cooper HS, Dawsey SM, Dixon MF, Fenoglio-Preiser CM, Flejou JF, Geboes K, Hattori T, Hirota T, Itabashi M, Iwafuchi M, Iwashita A, Kim YI, Kirchner T, Klimpfinger M, Koike M, Lauwers GY, Lewin KJ, Oberhuber G, Offner F, Price AB, Rubio CA, Shimizu M, Shimoda T, Sipponen P, Solcia E, Stolte M, Watanabe H, Yamabe H. The Vienna classification of gastrointestinal epithelial neoplasia. Gut. 2000 Aug;47(2):251-5. doi: 10.1136/gut.47.2.251. PMID 10896917
- [Background] Guo S, Diep D, Plongthongkum N, Fung HL, Zhang K, Zhang K. Identification of methylation haplotype blocks aids in deconvolution of heterogeneous tissue samples and tumor tissue-of-origin mapping from plasma DNA. Nat Genet. 2017 Apr;49(4):635-642. doi: 10.1038/ng.3805. Epub 2017 Mar 6. PMID 28263317
- [Background] Cai G, Cai M, Feng Z, Liu R, Liang L, Zhou P; ColonAiQ Group; Zhu B, Mo S, Wang H, Lan X, Cai S, Xu Y, Wang R, Dai W, Han L, Xiang W, Wang B, Guo W, Zhang L, Zhou C, Luo B, Li Y, Nie Y, Ma C, Su Z. A Multilocus Blood-Based Assay Targeting Circulating Tumor DNA Methylation Enables Early Detection and Early Relapse Prediction of Colorectal Cancer. Gastroenterology. 2021 Dec;161(6):2053-2056.e2. doi: 10.1053/j.gastro.2021.08.054. Epub 2021 Sep 4. No abstract available. PMID 34487783